CLINICAL TRIAL: NCT06295939
Title: Effect of Social Support Program on Grief of Pregnancy Loss in Sunpasitthiprasong Hospital: a Randomized Controlled Trial
Brief Title: Effect of Social Support Program on Grief of Pregnancy Loss in Sunpasitthiprasong Hospital
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanpasitthiprasong Hospital (Other Government)
Responsible Party: Principal Investigator, Adina Srisomboon, Principal Investigator, Sanpasitthiprasong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CA code 016/2565, 012/2566
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Loss; Grief; Social Support
Keywords: Pregnancy Loss; Grief and Loss; Social support program

STUDY DESIGN:
Intervention Model Description: 1. The researcher provided information about a research project involving pregnant women diagnosed with fetal demise or abnormalities, who are recommended to undergo pregnancy termination at the third trimester abortion clinic.
  2. Pregnant women voluntarily consent to participate in the research by signing the informed consent form.
  3. Volunteer participants providing consent will be randomly divided into two groups using the randomization technique with Excel program.
  4. Divide into groups of 45 individuals each, totaling 90 participants in the entire sample.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, the control group (Experimental): Group 1 the control group receive routine nursing care from the assigned nurse.
  Interventions: Other: Routine nursing care
- Group 2: the experimental group (Experimental): Group 2, the experimental group, will receive regular nursing care from the assigned nurse and a social support program provided by the researcher Phase 1 (Before Pregnancy Termination) Phase 2 (After Pregnancy Termination, Before Returning Home)
  Interventions: Other: social support program; Other: Routine nursing care

INTERVENTIONS:
Other: social support program — Group 2, the experimental group, will receive routine nursing care from the assigned nurse and a social support program provided by the researcher, as follows:
  Phase 1 (Before Pregnancy Termination)
  Phase 2 (After Pregnancy Termination, Before Returning Home):
  Arms: Group 2: the experimental group
Other: Routine nursing care — The sample group will receive routine nursing care from the assigned nurse.

SUMMARY:
Research Question:

Does participation in a social support program have an impact on the Perinatal Grief Scale of women who experience pregnancy loss through abortion? Research hypothesis

1. The grief scores from pregnancy loss among women who had to terminate their pregnancies in the group receiving social support program were lower than those in the group receiving standard nursing care.
2. The grief scores from pregnancy loss among women who had to terminate their pregnancies after receiving the social support program were lower than those before receiving the social support program.

Primary Objectives:

To study the grief and sorrow resulting from the loss of a fetus due to pregnancy termination in women who have undergone social support programs, in comparison to those who have received regular nursing care.

Secondary Objectives:

1. To investigate the grief and sorrow resulting from the loss of a fetus due to pregnancy termination after receiving social support programs compared to before receiving such programs.
2. To examine the grief and sorrow following pregnancy termination before returning home and one month after miscarriage.
3. To explore other outcomes of pregnancy termination, such as complete abortion, uterine curettage, and post-miscarriage complications.

DETAILED DESCRIPTION:
Research Methodology:

The research is a randomized controlled trial (RCT) of the single-blinded type. In this design, the evaluator, or research assistant, is unaware of the participants; group assignments, meaning they do not know which individuals belong to the experimental group and which ones belong to the control group.

Population and Sample:

Population: The population for this study comprises females who have undergone abortion and are admitted for post-abortion care at the obstetrics 3 wards in Sunpasitthiprasong hospital.

Sample: The sample for this study will be selected from the aforementioned population. The selection criteria for the sample are defined as follows:

1. Pregnant women diagnosed with fetal demise and requiring pregnancy termination.
2. Fetus with abnormalities requiring pregnancy termination.
3. Age between 18 and 45 years.
4. Gestational age not exceeding 24 weeks.
5. No history of mental illness.
6. No hearing, visual, speech impairments, and able to read and write in the Thai language.

Exclusion Criteria:

1. Pregnant women diagnosed with an ectopic pregnancy.
2. Presence of severe complications such as hemorrhage or shock.
3. Women undergoing a pregnancy termination due to criminal abortion.

Research Tools:

Experimental Tools

Social Support Program:

1.1 The social support program is developed based on the conceptual framework by House (1981) and is informed by relevant literature, textbooks, and research studies. The program is designed to provide support in two phases: Phase 1: Before the abortion procedure. Phase 2: After the abortion procedure. 1.2 Abortion Education Plan: The educational plan includes instructional content on abortion, methods of abortion, pain relief during abortion, post-abortion self-care, grief and loss, and coping with sadness.

1.3 Self-Care Manual for Women Undergoing Abortion: This manual encompasses guidance on abortion, abortion methods, pain relief during abortion, post-abortion self-care, dealing with grief, and grief management.

Data Collection Tools:

2.1 Personal Information and Pregnancy Data Questionnaire: A questionnaire capturing personal information and pregnancy-related data. Includes items such as age, marital status, occupation, education level, family income, healthcare entitlement, desire for children before diagnosis of fetal abnormality, gestational age at the time of abortion, abnormality leading to abortion, abortion method, duration of the abortion procedure, completeness of the abortion, and complications arising from the abortion.

2.2 Perinatal Grief Assessment Questionnaire (Perinatal Grief Scale short version - PGS-33): This questionnaire, translated into Thai by Sukanya Kritiyutanon (2014) and adjusted based on expert suggestions, comprises 33 questions. It evaluates grief on three dimensions: Active grief, Difficulty coping, and Despair. Each question is rated on a 5-point Likert scale (Strongly Agree to Strongly Disagree), with scores ranging from 33 to 165. The higher the score, the higher the level of grief. Scores above 91 indicate a high level of grief.

Data Collection:

1. The researcher provided information about a research project involving pregnant women diagnosed with fetal demise or abnormalities, who are recommended to undergo pregnancy termination at the third trimester abortion clinic.
2. Pregnant women voluntarily consent to participate in the research by signing the informed consent form.
3. Volunteer participants providing consent will be randomly divided into two groups using the randomization technique with Excel program.
4. Divide into groups of 45 individuals each, totaling 90 participants in the entire sample.

   Group 1, the control group: Researchers will meet with the sample group on the first day of their stay at the patient care center. Participants will respond to personal information and a questionnaire assessing grief from pregnancy loss. Subsequently, the sample group will receive routine nursing care from the assigned nurse, who will explain the treatment plan provided by the physician, follow the physician's treatment orders, and provide post-abortion care. On the morning of that day, the research assistant, a nurse from obstetrics 3 ward on duty, will visit the sample group to administer the grief assessment questionnaire.

   Group 2, the experimental group, will receive routine nursing care from the assigned nurse and a social support program provided by the researcher, as follows:

   Phase 1 (Before Pregnancy Termination): On the first day of their stay at the hospital, the researcher will meet with the sample group. Participants will respond to a general information questionnaire and an assessment of grief from pregnancy loss. Subsequently, the sample group will receive nursing care according to the social support program. The researcher will establish rapport, provide information about the reasons for pregnancy termination, explain the steps of the procedure, discuss potential symptoms after termination, teach pain management techniques during the procedure, and engage in supportive conversations. This session will last approximately 30 minutes.

   Phase 2 (After Pregnancy Termination, Before Returning Home): Before leaving the hospital, the researcher will provide information about potential post-abortion symptoms, such as mild abdominal pain that may gradually subside, a gradual decrease in vaginal bleeding within 1-2 weeks, and instructions to seek medical attention if bleeding persists, there is a foul smell, or if the patient develops a fever. The researcher will also offer knowledge about grief, provide emotional support, and discuss self-care after pregnancy termination. Additionally, information will be given about preparing for future pregnancies. This session will take about 30 minutes. A follow-up appointment will be scheduled for a post-abortion checkup with the nurse from obstetrics 3 ward on duty on the same morning, who will administer the grief assessment questionnaire.
5. The researcher scheduled appointments for both the control and experimental groups on the same day as the post-abortion checkup with the physician (1 month after pregnancy termination). The research assistant administered the grief assessment questionnaire to both the control and experimental groups during this follow-up appointment.
6. The researcher recorded pregnancy, childbirth, and outcomes of pregnancy termination data, including the desire for pregnancy before diagnosis of fetal abnormalities, gestational age at the time of pregnancy termination, fetal abnormalities leading to termination, termination methods, duration of the termination procedure, completeness of abortion, the use of dilation and curettage, and complications resulting from pregnancy termination.

The duration of hospital stay could not be specified and depended on the physician's treatment plan but typically did not exceed 24-48 hours after completing the abortion

Data collection and management include a Questionnaire and The researcher analyzed the data using the SPSS version 25.0 statistical.

1. Descriptive Data Analysis: Descriptive statistics, including counts (percentages), mean, standard deviation (SD), median, and interquartile range,
2. Comparison of Depression Scores between Control and Experimental Groups after Receiving the Program: Independent t-test and Mann-Whitney U test were utilized for normally distributed and non-normally distributed data, respectively.
3. Comparison of Depression Scores before and after Program Implementation: Paired t-test was employed to compare depression scores before and after the program.
4. Comparison of Categorical Data: Chi-square test and Fisher's exact test were used for analyzing count data.
5. Intention-to-Treat Analysis: The intention-to-treat principle was applied, considering a statistical significance level of .05

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women diagnosed with fetal demise and requiring pregnancy termination.
2. Fetus with abnormalities requiring pregnancy termination.
3. Age between 18 and 45 years.
4. Gestational age not exceeding 24 weeks.
5. No history of mental illness.
6. No hearing, visual, speech impairments, and able to read and write in the Thai language.

Exclusion Criteria:

1. Pregnant women diagnosed with an ectopic pregnancy.
2. Presence of severe complications such as hemorrhage or shock.
3. Women undergoing a pregnancy termination due to criminal abortion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The Perinatal Grief Assessment Questionnaire. | 1 month
  The Perinatal Grief Assessment Questionnaire (Perinatal Grief Scale short version - PGS-33):
  This questionnaire, translated into Thai by Sukanya Kritiyutanon (2014) and adjusted based on expert suggestions, comprises 33 questions. It evaluates grief on three dimensions: Active grief, Difficulty coping, and Despair. Each question is rated on a 5-point Likert scale (Strongly Agree to Strongly Disagree), with scores ranging from 33 to 165. The higher the score, the higher the level of grief. Scores above 91 indicate a high level of grief.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanpasitthiprasong Hospital, Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: No